CLINICAL TRIAL: NCT06298175
Title: Self-Management Training With Online Intervention Process for Young Adults With Chronic Conditions: Effects on Self-Management, Emotion Regulation, and Occupational Balance: A Randomized Controlled Study
Brief Title: Self-Management Training With Online Intervention Process for Young Adults With Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Esma Ozkan, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-157
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Chronic Disease
Keywords: Self-Management; Chronic Conditions; Young Adults
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Pre-post test, randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The study group received 8 weeks of self-management training. Reflections, prepared using Power Point, were used in all sessions. The study employed various methods, including the question-answer and audio-visual methods, as well as performance feedback when necessary during the sessions. Final evaluations were conducted for both groups after eight weeks.
  Interventions: Behavioral: Self management training
- Control Group (Active Comparator): The control group was informed about self-management for 1 week. General information was given about approaches to improving self-management. Final evaluations were conducted for both groups after eight weeks.
  Interventions: Behavioral: Self management training

INTERVENTIONS:
Behavioral: Self management training — The self-management training programme for the study group consisted of eight sessions. Each session lasted between 40 and 50 minutes and followed a structured format: a 5-minute introduction, a 5-minute summary of the previous session, and a 30-40 minute presentation on the session's topic. Training plan on cognition, emotion regulation and self-management was implemented

SUMMARY:
The study was conducted from 15th April 2021 to 15th August 2021. It employed a pretest-posttest design with control and training groups. In this study, a pretest-posttest design including control and training groups was used. Pre-assessments were taken from young adults who reported that they wanted to participate in the study via social media accounts and e-mail and who met the study criteria, and two groups were formed by the simple randomization method. The study group received 8 weeks of self-management training. The control group was informed about self-management for 1 week. Final evaluations were conducted for both groups after eight weeks.

DETAILED DESCRIPTION:
Pre-assessments were taken from young adults who reported that they wanted to participate in the study via social media accounts and e-mail and who met the study criteria, and two groups were formed by simple randomization method. The study group received 8 weeks of self-management training. The control group was informed about self-management for 1 week. Final evaluations were conducted for both groups after eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* having no communication barriers
* having a chronic disease such as asthma, diabetes, heart disease, or hypertension

Exclusion Criteria:

* being under 35 years old
* undergoing concurrent psychological treatment/therapy
* having Covid-19
* requiring treatment for other diseases during the training process

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Self-Control Self-Management Scale (SCMS) | pre-treatment and post-treatment up to 8-weeks
  The Self-Control and Self-Management Scale consists of three subscales: self-monitoring, self-evaluation and self-reinforcement. It is a 6-point Likert-type scale consisting of 16 items (0= Does not define me at all, 5= Defines me completely).

SECONDARY OUTCOMES:
Cognitive Emotion Regulation Questionnaire (CERQ) | pre-treatment and post-treatment up to 8-weeks
  The five-point Likert-type scale (1 = not at all suitable for me, 2 = somewhat suitable for me, 3 = partially suitable for me, 4 = very suitable for me, 5 = completely suitable for me) consists of a total of 36 items. It consists of nine sub-dimensions: self-blame, acceptance, rumination, positive refocusing, refocus on planning, positive reappraisal, putting into perspective, catastrophizing, and other-blame.
The Occupational Balance Questionnaire (OBQ) | pre-treatment and post-treatment up to 8-weeks
  In 2019, Günal et al. conducted a validity and reliability study of the 11-item revised version of the questionnaire in Turkish. The scale consists of four response categories (strongly disagree, disagree, agree, strongly agree), with each item being assigned a value between 0 and 3 points. The sum of the individual items results in a score between 0 and 33.

CONTACTS AND LOCATIONS:
Overall Officials: Esma Ozkan, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No